CLINICAL TRIAL: NCT06366542
Title: The Effect of Using Virtual Reality on Balance in People With Persistent Postural-Perceptual Dizziness
Brief Title: Virtual Reality in People With Persistent Postural-Perceptual Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2024
Record Dates: First submitted 2024-03-25; First posted 2024-04-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Vestibular Dizziness
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Therapy (VRT) (Active Comparator): Participants went through conventional VRT in addition to optokinetic exercise training. The VRT exercises were composed of gaze stabilization, head motion, and postural stability exercises with static and dynamic balance exercises. Ten repetitions of each VRT exercise were practiced in the same session for three sets. Moreover, participants were instructed to watch optokinetic stimulation videos. The optokinetic stimulation training was conducted using the following displays (a mobile and TV screen).
  Interventions: Other: Vestibular Rehabilitation Therapy (VRT); Other: Optokinetic Stimulation exercises
- Virtual Reality (Experimental): The same intervention program for the control group was implemented for participants in the experimental group, with the addition of using the VR split screen in Samsung Gear VR goggles in the last 4 sessions. Using the VR goggles, participants started watching the videos for 30 seconds to 1 minute in the sitting position in the first two sessions, followed by 1-2 minutes in the standing position for the last 2 sessions.
  Interventions: Other: Vestibular Rehabilitation Therapy (VRT); Other: Virtual reality exercises; Other: Optokinetic Stimulation exercises

INTERVENTIONS:
Other: Vestibular Rehabilitation Therapy (VRT) — The VRT exercises were composed of gaze stabilization, head motion and postural stability exercises with static and dynamic balance exercises.
  Other Names: VRT
Other: Virtual reality exercises — The VR exercises included watching theraputic videos using the virtual reality goggles with static and dynamic balance exercises.
  Other Names: VR
  Arms: Virtual Reality
Other: Optokinetic Stimulation exercises — Optokinetic Stimulation is a type of visual stimulation used to improve visual function and balance in patients with vestibular disorders.

SUMMARY:
This study aimed to compare the effectiveness of virtual reality (VR) and vestibular rehabilitation therapy (VRT) in enhancing balance in individuals with Persistent Postural-Perceptual Dizziness (PPPD). The experimental group received VR combined with VRT and optokinetic stimulation, while the control group received VRT and optokinetic stimulation. The study involved 42 individuals diagnosed with PPPD and administered ten intervention sessions over six weeks. The study also examined the impact of VR on various aspects of PPPD, including dizziness, visual vertigo, mental well-being, sleep quality, fall risk, and overall quality of life.

DETAILED DESCRIPTION:
Persistent Postural-Perceptual Dizziness (PPPD) represents a relatively new vestibular diagnosis that has garnered recent attention within the medical community. Consequently, there exists a pressing demand for efficacious and innovative management strategies. The primary purpose of this study was to assess the comparative effectiveness of virtual reality (VR) versus vestibular rehabilitation therapy (VRT) in enhancing balance among individuals afflicted with PPPD. A secondary purpose encompassed an investigation of VR's impact on various dimensions of PPPD, including dizziness, visual vertigo, mental well-being, sleep quality, fall risk, and overall quality of life. Materials and Methods: A cohort comprising forty-two individuals conclusively diagnosed with PPPD was randomly assigned to two distinct groups. The experimental cohort comprised twenty-one participants subjected to a combination of VR with optokinetic stimulation alongside VRT, whereas the control group, also consisting of twenty-one individuals, underwent solely optokinetic stimulation paired with VRT. The intervention sessions were administered twice weekly over a span of six weeks, resulting in a total of ten intervention sessions. Additionally, baseline and post-intervention assessments were conducted to gauge the efficacy of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of the PPPD from a specialized physician, based on the diagnostic criteria published by the Barany Society.
* Patients who scored more than 27 on the Niigata PPPD Questionnaire (NPQ)

Exclusion Criteria:

* If they suffered from other neurological or orthopedic deficits that affected their balance and prevented them from moving independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Niigata Persistent Postural-Perceptual Dizziness Questionnaire (NPQ) | Before intervention.
  self-reported questionnaire that was generated to screen for and assess the severity of Persistent Postural-Perceptual Dizziness. Higher score is worse severity of Persistent Postural-Perceptual Dizziness. Minimum score is 0 and maximum score is 72.
The Niigata Persistent Postural-Perceptual Dizziness Questionnaire (NPQ) | After 6 weeks
  self-reported questionnaire that was generated to screen for and assess the severity of Persistent Postural-Perceptual Dizziness. Higher score is worse severity of Persistent Postural-Perceptual Dizziness. Minimum score is 0 and maximum score is 72.
The Niigata Persistent Postural-Perceptual Dizziness Questionnaire (NPQ) | After one year follow up.
  self-reported questionnaire that was generated to screen for and assess the severity of Persistent Postural-Perceptual Dizziness. Higher score is worse severity of Persistent Postural-Perceptual Dizziness. Minimum score is 0 and maximum score is 72.
Dizziness Handicap Inventory (DHI) | Before intervention.
  self- reported questionnaire that assesses the perceived disability from dizziness. Higher score indicates worse disability from dizziness. Minimum score is 0 and maximum score is 100.
Dizziness Handicap Inventory (DHI) | After 6 weeks
  self- reported questionnaire that assesses the perceived disability from dizziness. Higher score indicates worse disability from dizziness. Minimum score is 0 and maximum score is 100.
Falls Efficacy Scale International (FES-I) | Before intervention.
  self-reported questionnaire that assesses fear of falling. A higher score means worse concerns from falling. Minimum score is 16 and maximum score is 64.
Falls Efficacy Scale International (FES-I) | After 6 weeks
  self-reported questionnaire that assesses fear of falling. A higher score means worse concerns from falling. Minimum score is 16 and maximum score is 64.
Dynamic Gait Index (DGI) | Before intervention.
  A clinical performance-based tool that is used to evaluate dynamic postural stability. A higher score indicates better dynamic balance and gait. Minimum score is 0 and maximum score is 24.
Dynamic Gait Index (DGI) | After 6 weeks
  A clinical performance-based tool that is used to evaluate dynamic postural stability. A higher score indicates better dynamic balance and gait. Minimum score is 0 and maximum score is 24.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Before intervention.
  A self-reported questionnaire that assesses quality of sleep. A higher score indicates worse sleep quality. Minimum score is 0 and maximum score is 21.
Pittsburgh Sleep Quality Index (PSQI) | After 6 weeks
  A self-reported questionnaire that assesses quality of sleep. A higher score indicates worse sleep quality. Minimum score is 0 and maximum score is 21.
Hospital Anxiety and Depression Scale (HADS) | Before intervention.
  a self-assessment scale that was developed to assess the severity of mood disturbances including depression and anxiety. Higher scores mean worse severity in depression and anxiety. Minimum score is 0 and maximum score is 21 for each subscale (depression and anxiety).
Hospital Anxiety and Depression Scale (HADS) | After 6 weeks
  a self-assessment scale that was developed to assess the severity of mood disturbances including depression and anxiety. Higher scores mean worse severity in depression and anxiety. Minimum score is 0 and maximum score is 21 for each subscale (depression and anxiety).
Medical Outcomes Study Short Form 12 (SF-12) | Before intervention.
  A self-reported questionnaire that assesses the impact of any health condition on the quality of life. Higher scores indicate better quality of life. Minimum score is 0 and maximum score is 100.
Medical Outcomes Study Short Form 12 (SF-12) | After 6 weeks
  A self-reported questionnaire that assesses the impact of any health condition on the quality of life. Higher scores indicate better quality of life. Minimum score is 0 and maximum score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Alia A Alghwiri, PhD, Principal Investigator — The University of Jordan
Locations (1):
- Royal Medical Services, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.